CLINICAL TRIAL: NCT06884332
Title: Étude de Non infériorité Sur l'Impact de la Diminution Des Volumes d'Irradiations vertébraux en Cas d'Irradiation Palliative Rachidienne métastatique Osseuse Sur l'efficacité Antalgique
Brief Title: Spinal Palliation in Irradiation for Neoplastic Analgesia and Life Quality
Acronym: SPINAL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut de Cancérologie de Lorraine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024-A02789-38
Record Dates: First submitted 2025-03-03; First posted 2025-03-19 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Bone Metastasis; Oncology Pain
Keywords: Bone metastasis; Irradiation; Palliative; Analgesic
MeSH Terms: conditions — Cancer Pain

STUDY DESIGN:
Intervention Model Description: This is a prospective, phase III, multicenter, non-inferiority, randomized (1:1) therapeutic clinical trial with two arms, evaluating the efficacy and tolerance of targeted analgesic irradiation limited to the affected vertebrae.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional spinal irradiation (Active Comparator): Spinal irradiation without sparing the adjacent vertebrae.
  Interventions: Radiation: Conventional spinal irradiation
- Sparing irradiation (Experimental): Spinal irradiation while sparing the adjacent vertebrae.
  Interventions: Radiation: Sparing irradiation

INTERVENTIONS:
Radiation: Sparing irradiation — For "Sparing irradiation" arm the Clinical Target Volume (CTV) = Growth Tumor Volume (GTV) + entire vertebra opposite.
  Arms: Sparing irradiation
Radiation: Conventional spinal irradiation — For "conventional spinal irradiation" arm, Clinical Target Volume (CTV ) = Growth Tumor Volume (GTV) + entire vertebra opposite + 1 vertebra above and below.
  Arms: Conventional spinal irradiation

SUMMARY:
The goal of this clinical trial is to assess the impact of reducing the volume of palliative metastatic bone irradiation on analgesic effectiveness at day 30 and to evaluate the efficiency of telemonitoring in identifying patients who could benefit from Patient-Reported Outcomes (PROs) and require care.

These objectives will be addressed in a multicenter, randomized, prospective study with two arms:

A standard arm with spinal irradiation without sparing the adjacent vertebrae. An experimental arm with spinal irradiation sparing the adjacent vertebrae. The results will determine whether reducing the irradiated volume can maintain effective pain relief while minimizing side effects.

DETAILED DESCRIPTION:
Palliative analgesic radiotherapy (RT) is used to relieve pain in patients with bone metastases. This technique involves irradiating the vertebrae above and below the ones responsible for the pain. Traditional two-dimensional radiotherapy (2D-RT) was characterized by a physical penumbra that could extend up to 50% of a vertebra's height, leading to underdosing of the target volume and, consequently, reduced analgesic effectiveness.

However, computed tomography (CT) scans or CT-based imaging have replaced these practices, allowing for high precision in delineating target volumes. Despite advancements in irradiation techniques, the physical penumbra is now negligible with modern machines, reducing the need for large margins and thereby limiting side effects associated with the irradiation of healthy tissues.

These factors have led us to conduct a clinical trial to assess the impact of reducing the volume of palliative metastatic bone irradiation on analgesic effectiveness at day 30 (D30) and to evaluate the efficiency of telemonitoring in identifying patients who could benefit from Patient-PROs and require care.

These objectives will be pursued in a multicenter, randomized, prospective study with two arms:

A standard arm, with spinal irradiation without sparing the adjacent vertebrae. An experimental arm, with spinal irradiation sparing the adjacent vertebrae. The results will determine whether reducing the irradiated volume can maintain effective pain relief while minimizing side effects. This could lead to changes in current palliative radiotherapy practices, reduce toxicity risks, and improve patients' quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Patient with bone pain related to at least 1 or more bone metastases of spinal location, contiguous or not, cervical (excluding C1), thoracic, lumbar or sacral up to and including S2; a patient can be included even if he or she is irradiated concomitantly or not for analgesic purposes on another non-spinal bone metastatic site. Bone lesions are objective on an imaging examination less than 3 months old: CT and/or MRI and/or PET and/or bone scintigraphy;
* Patient with at least moderate pain with EN ≥ 5;
* Patient on analgesic drug treatment for at least 7 days or poor tolerance of analgesics;
* Patient irradiated for palliative analgesic purposes. Post-cementoplasty irradiation is possible; an extension to the soft tissues is not a contraindication to inclusion;
* Patient with a validated palliative bone irradiation plan: 8 Gy / 1 fr or 20 Gy / 5 fr;
* Patient with planning only in static IMRT, arc therapy or helical tomotherapy;
* Patient with a primary cancer or a haemopathy;
* Patient currently undergoing or not a specific oncological systemic treatment, left to the discretion of the investigating physician;
* Patient currently undergoing or not a treatment with bisphosphonates and denosumab, left to the discretion of the investigating physician;
* WHO ≤ 2;
* Patient with a life expectancy ≥ 3 months;
* Patient able and agreeing to follow all study procedures in accordance with the protocol;
* Patient having understood, signed and dated the consent form;
* Patient affiliated to the social security system.

Exclusion Criteria:

* Pediatric patient;
* Patient undergoing stereotaxic irradiation;
* Patient undergoing oligometastatic disease;
* Patient undergoing re-irradiation unless the dose is not limiting to OARs;
* Patient treated with RT2D (conventional 2-dimensional radiotherapy) or RT3D (conventional 3-dimensional radiotherapy);
* Patient with MESCC (metastatic epidural spinal cord compression) except for a Bilsky grade < 1b;
* Patient who does not have a means of responding to online questionnaires;
* Patient and their entourage who cannot read or express themselves in French;
* Visually impaired patient;
* Patient already included in another therapeutic trial with an experimental molecule;
* Persons deprived of liberty or under guardianship (including curatorship).
* Pregnant woman, likely to be pregnant, or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 598 (Estimated)
Dates: Start 2025-07-02 (Actual); Primary Completion 2027-07-02 (Estimated); Study Completion 2029-01-02 (Estimated)

PRIMARY OUTCOMES:
Impact of Reducing the Volume of Palliative Bone Metastatic Irradiation on Analgesic Efficacy | From enrollment to the end of treatment at day 30 after the first irradiation.
  Pain response at day 30 at the site of the irradiated lesion will be assessed according to the international consensus definitions on bone metastases, using a numerical scale (0 to 10) and the consumption of equivalent opioids.

SECONDARY OUTCOMES:
Tolerance of Reducing the Volume of Palliative Bone Metastatic Irradiation | From enrollment to the 30 days after the first irradiation session
  Tolerance will be assessed by the occurrence of toxicities according to the National Cancer Institute (NCI) PRO-Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.
Impact of a remote monitoring tool on quality of life | From enrollment to the 30 days after the first irradiation session
  Quality of life will be assessed using questionnaire EORTC QLQ-C15PAL ; the score scale is from 0 to 100.
Evaluation of Quality of life Bone Metastases Module | From enrollment to the 30 days after the first irradiation session
  Quality of life will be assessed using questionnaires EORTC QLQ-Bone Metastases (BM)22. The score scale ranges from 0 to 100.
Level of adherence | From enrollment to 45 days after the first irradiation
  The level of adherence will be assessed based on the rate of compliance with completing the online questionnaires by the patient or their caregivers. The score scale ranges from 0 to 100.
Use of a remote monitoring tool | From enrollment to 45 days after the first irradiation
  The handling of the digital tool will be assessed by the System Usability Scale (SUS).The score scale ranges from 0 to 100.
Patient satisfaction | From enrollment to 30 months after the first irradiation
  Patient satisfaction will be measured according to the PACIC (Patient Assessment Chronic Illness Care) score. The total score ranges from 1 to 5.
Medical care patient satisfaction | From enrollment to 30 months after the first irradiation.
  Patient satisfaction will be measured according the questionnaire concerning medical care (PEC). The score scale ranges from 0 to 100.
Rate of analgesic re-irradiation | From enrollment to 30 days after the first irradiation session and after 12 months
  The administration of a supplementary dose of irradiation between Day 30 and Month 12 will be recorded
Correlation between dosimetric constraints for organs at risk (OARs) and the associated grade 0, 1, 2, and 3 acute toxicities | From enrollment to 12 months after the first irradiation session.
  Doses to OARs will be collected for the main organs at risk (OARs) in the vicinity by exporting the dose-volume histograms for each organ at risk.
Construction of a Prognostic Score | From enrollment to 12 months after the first irradiation session.
  A prognostic score will be constructed from the variables of all the prognostic factors collected in this study. The score scale ranges from 0 to 100.
Overall survival | From enrollment to 12 months after the first irradiation session.
  Overall survival will be calculated as the time elapsed between the end of treatment and the date of death, from all causes.

CONTACTS AND LOCATIONS:
Overall Officials: Nour MAMMARI HALABI, PhD., Study Chair — Institut de Cancérologie de Lorraine
Locations (4):
- France (4):
  - Centre Hospitalier Universitaire de Brest, Brest, Brest
  - Centre Henri Becquerel Rouen, Rouen, Rouen
  - Institut de cancérologie de l'Ouest (ICO), Saint-Herblain, Saint-Herblain
  - Institut de Cancérologie de Lorraine, Vandœuvre-lès-Nancy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Temel JS, Greer JA, Muzikansky A, Gallagher ER, Admane S, Jackson VA, Dahlin CM, Blinderman CD, Jacobsen J, Pirl WF, Billings JA, Lynch TJ. Early palliative care for patients with metastatic non-small-cell lung cancer. N Engl J Med. 2010 Aug 19;363(8):733-42. doi: 10.1056/NEJMoa1000678. PMID 20818875
- [Background] Fisher CG, DiPaola CP, Ryken TC, Bilsky MH, Shaffrey CI, Berven SH, Harrop JS, Fehlings MG, Boriani S, Chou D, Schmidt MH, Polly DW, Biagini R, Burch S, Dekutoski MB, Ganju A, Gerszten PC, Gokaslan ZL, Groff MW, Liebsch NJ, Mendel E, Okuno SH, Patel S, Rhines LD, Rose PS, Sciubba DM, Sundaresan N, Tomita K, Varga PP, Vialle LR, Vrionis FD, Yamada Y, Fourney DR. A novel classification system for spinal instability in neoplastic disease: an evidence-based approach and expert consensus from the Spine Oncology Study Group. Spine (Phila Pa 1976). 2010 Oct 15;35(22):E1221-9. doi: 10.1097/BRS.0b013e3181e16ae2. PMID 20562730
- [Background] Basch E, Barbera L, Kerrigan CL, Velikova G. Implementation of Patient-Reported Outcomes in Routine Medical Care. Am Soc Clin Oncol Educ Book. 2018 May 23;38:122-134. doi: 10.1200/EDBK_200383. PMID 30231381
- [Background] Marino D, Baratelli C, Guida G, Turco CGC, Lacidogna G, Sperti E, Vignani F, De Luca E, Zichi C, Audisio M, Ballaminut D, Bellezza A, Chiotto P, Ciriolo G, Comite R, Codegone F, Florio S, Fusco L, Polimeno L, Pozzi D, Zilio E, Terzolo S, Di Maio M. Impact of adoption of patient-reported outcomes in clinical practice on the accuracy of symptom reporting in medical records of cancer patients. Recenti Prog Med. 2020 Dec;111(12):740-748. doi: 10.1701/3509.34965. PMID 33362171
- [Background] Basch E, Iasonos A, McDonough T, Barz A, Culkin A, Kris MG, Scher HI, Schrag D. Patient versus clinician symptom reporting using the National Cancer Institute Common Terminology Criteria for Adverse Events: results of a questionnaire-based study. Lancet Oncol. 2006 Nov;7(11):903-9. doi: 10.1016/S1470-2045(06)70910-X. PMID 17081915
- [Background] Di Maio M, Gallo C, Leighl NB, Piccirillo MC, Daniele G, Nuzzo F, Gridelli C, Gebbia V, Ciardiello F, De Placido S, Ceribelli A, Favaretto AG, de Matteis A, Feld R, Butts C, Bryce J, Signoriello S, Morabito A, Rocco G, Perrone F. Symptomatic toxicities experienced during anticancer treatment: agreement between patient and physician reporting in three randomized trials. J Clin Oncol. 2015 Mar 10;33(8):910-5. doi: 10.1200/JCO.2014.57.9334. Epub 2015 Jan 26. PMID 25624439
- [Background] Stromgren AS, Groenvold M, Sorensen A, Andersen L. Symptom recognition in advanced cancer. A comparison of nursing records against patient self-rating. Acta Anaesthesiol Scand. 2001 Oct;45(9):1080-5. doi: 10.1034/j.1399-6576.2001.450905.x. PMID 11683656
- [Background] Basch E. The missing voice of patients in drug-safety reporting. N Engl J Med. 2010 Mar 11;362(10):865-9. doi: 10.1056/NEJMp0911494. No abstract available. PMID 20220181
- [Background] Del Gaudio AC, Carpenter PJ, Stein LS, Morrow G. Characteristics of patients completing referrals from an emergency department to a psychiatric outpatient clinic. Compr Psychiatry. 1977 May-Jun;18(3):301-7. doi: 10.1016/0010-440x(77)90026-8. No abstract available. PMID 858248
- [Background] Klish DS, Grossman P, Allen PK, Rhines LD, Chang EL. Irradiation of spinal metastases: should we continue to include one uninvolved vertebral body above and below in the radiation field? Int J Radiat Oncol Biol Phys. 2011 Dec 1;81(5):1495-9. doi: 10.1016/j.ijrobp.2010.07.2007. Epub 2010 Nov 11. PMID 21074335
- [Background] Alcorn S, Cortes AA, Bradfield L, Brennan M, Dennis K, Diaz DA, Doung YC, Elmore S, Hertan L, Johnstone C, Jones J, Larrier N, Lo SS, Nguyen QN, Tseng YD, Yerramilli D, Zaky S, Balboni T. External Beam Radiation Therapy for Palliation of Symptomatic Bone Metastases: An ASTRO Clinical Practice Guideline. Pract Radiat Oncol. 2024 Sep-Oct;14(5):377-397. doi: 10.1016/j.prro.2024.04.018. Epub 2024 May 22. PMID 38788923
- [Background] van der Velden J, Willmann J, Spalek M, Oldenburger E, Brown S, Kazmierska J, Andratschke N, Menten J, van der Linden Y, Hoskin P. ESTRO ACROP guidelines for external beam radiotherapy of patients with uncomplicated bone metastases. Radiother Oncol. 2022 Aug;173:197-206. doi: 10.1016/j.radonc.2022.05.024. Epub 2022 May 31. PMID 35661676
- [Background] Chow E, Hoskin P, Mitera G, Zeng L, Lutz S, Roos D, Hahn C, van der Linden Y, Hartsell W, Kumar E; International Bone Metastases Consensus Working Party. Update of the international consensus on palliative radiotherapy endpoints for future clinical trials in bone metastases. Int J Radiat Oncol Biol Phys. 2012 Apr 1;82(5):1730-7. doi: 10.1016/j.ijrobp.2011.02.008. Epub 2011 Apr 12. PMID 21489705